CLINICAL TRIAL: NCT06082908
Title: Predictors of the Disability in Nursing Home Residents: a Descriptive Study
Brief Title: Geriatric Syndrome in Nursing Home Residents
Status: Completed | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Ulkukezbansahin, Assistant Professor in Department of Therapy and Rehabilitation, Giresun University
Other Study IDs: Nursing home
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2023-10

CONDITIONS: Disability Physical
Keywords: geriatric assessment; activities of daily living; nutritional deficiency; functional dependence; urinary incontinence
MeSH Terms: conditions — Malnutrition; Urinary Incontinence | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Diagnostic test — Subjective and objective measurement will be performed in older adults.

SUMMARY:
Disability in daily living activities (ADL) is a typical issue among nursing care residents. The goal of this study was to look at the geriatric syndromes that cause incapacity in nursing home residents.

DETAILED DESCRIPTION:
More often than not, people who live in nursing homes can't move out. One of the main reasons they leave their own home is to lose their freedom. Nursing homes also have a lot of people with geriatric diseases like cognitive impairment, balance problems, urinary incontinence, and disability. But it's not known what role geriatric syndromes play in ADL impairment. To come up with good ways to treat geriatric syndromes, which are the main causes of ADL disability in nursing home patients, we need to know more about them. So, the point of this study was to look into geriatric syndromes that are linked to disability and find out what causes disability in nursing home patients.

ELIGIBILITY:
Inclusion Criteria:

* age over 65
* staying in a nursing home for at least 12 months
* consent to participate in the study were the inclusion criteria.

Exclusion Criteria:

* people who were mentally unable to answer questions,
* people who were hospitalized
* people who had severe hearing or vision problems that made it hard to communicate
* people who took benzodiazepines or psychotropic drugs that made it hard to walk or balance
* people who had fractures or endoprostheses in any part of their bodies.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This cross-sectional study was conducted in nursing homes located in two cities.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
frailty | 5 minute
  FRAIL includes five items that evaluate ambulation, weight loss, fatigue, diseases, and resistance.
  Each item receives a value of 0 or 1, for a total score ranging from 0 (best) to 5 (worst). A score of 3 shows frailty, a score of 1-2 indicates prefrailty, and a score of 0 indicates robustness.
disability | 5 minute
  The Barthel Index (BI) was used to determine the level of disability in ADL. The indicator has a maximum total score of 100, indicating that the individual is entirely autonomous in all physical functions. The lowest possible score is 0; this indicates that the individual is entirely dependent.

SECONDARY OUTCOMES:
sarcopenia | 5 minute
  The SARC-F questionnaire was used to assess the risk of sarcopenia. The indicator has a maximum total score of 100, indicating that the individual is entirely autonomous in all physical functions. The lowest possible score is 0; this indicates that the individual is entirely dependent.

CONTACTS AND LOCATIONS:
Overall Officials: ULKU K SAHIN, PhD, Principal Investigator — Giresun University
Locations (1):
- Giresun University, Giresun, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Vermeulen J, Neyens JC, van Rossum E, Spreeuwenberg MD, de Witte LP. Predicting ADL disability in community-dwelling elderly people using physical frailty indicators: a systematic review. BMC Geriatr. 2011 Jul 1;11:33. doi: 10.1186/1471-2318-11-33. PMID 21722355
- [Background] Jenkins KR, Fultz NH. Functional impairment as a risk factor for urinary incontinence among older Americans. Neurourol Urodyn. 2005;24(1):51-5. doi: 10.1002/nau.20089. PMID 15578629